CLINICAL TRIAL: NCT00000190
Title: Cocaine in Parotid Saliva, Blood and Urine
Brief Title: Cocaine in Parotid Saliva, Blood and Urine - 4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, James Cornish, Principal Investigator, University of Pennsylvania
Purpose: Diagnostic
Other Study IDs: NIDA-00144-4; 3R01DA012268 (NIH); K20-00144-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Detection; Parotid Saliva
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — parotid gland hypocalcemic protein, Bos taurus

INTERVENTIONS:
Procedure: Parotid Gland

SUMMARY:
The purpose of this study is to establish the use of parotid saliva as a means of detecting and quantifying cocaine and its metabolites.

ELIGIBILITY:
Please contact site for information.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 1991-01; Primary Completion 1992-02 (Actual); Study Completion 1992-02 (Actual)

PRIMARY OUTCOMES:
Cocaine & benzoylecgonine content in saliva, plasma, & urine

CONTACTS AND LOCATIONS:
Overall Officials: James Cornish, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States